CLINICAL TRIAL: NCT00745953
Title: Regression of Fatty Heart by Valsartan Therapy
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Dr. Ildiko Lingvay, MD, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IIRP Study US 73
Record Dates: First submitted 2008-08-29; First posted 2008-09-03 (Estimated); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Metabolic Syndrome; Lipotoxicity
Keywords: Metabolic syndrome; Lipotoxicity; Insulin sensitivity; Myocardial triglyceride levels; Hepatic triglyceride levels; Magnetic resonance spectroscopy
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance | interventions — Valsartan; Hydrochlorothiazide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Valsartan (Active Comparator): This arm will determine if blockade of the renin-angiotensin system reduces myocardial fat levels and improves insulin sensitivity. It consists of 6 visits: visit1 (baseline); visit2 (2 weeks); visit3 (1 month); visit4 (3 month); visit5 (6 month); visit6 (8 month). Visits 1 & 6 will consist of blood tests, glucose tolerance test by FSivGTT, MRS, & 24 hr ambulatory blood pressure monitoring. During visit 1, patients receive automatic blood pressure monitor, OMRON, to record blood pressure between visits. Visits 2 & 3 are needed for the adjustment of medication to the final dose level. During visits 4 & 5, Dr. Price will check subject's status as they continue the medication. In case of uncontrolled blood pressure, Dr. Price will prescribe amlodipine for the additional BP control.
  Interventions: Drug: Valsartan
- Hydrochlorothiazide (Active Comparator): This arm will determine if thiazide diuretics elevate myocardial triglyceride levels. It consists of 6 visits: visit1 (baseline); visit2 (2 weeks); visit3 (1 month); visit4 (3 month); visit5 (6 month); visit6 (8 month). Visits 1 & 6 will consist of blood tests, glucose tolerance test by FSivGTT, MRS, & 24 hr ambulatory blood pressure monitoring. During visit 1, patients receive automatic blood pressure monitor, OMRON, to record blood pressure between visits. Visits 2 & 3 are needed for the adjustment of medication to the final dose level. During visits 4 & 5, Dr. Price will check subject's status as they continue the medication. In case of uncontrolled blood pressure, Dr. Price will prescribe amlodipine for the additional BP control.
  Interventions: Drug: Hydrochlorothiazide

INTERVENTIONS:
Drug: Valsartan — Valsartan 320mg PO daily for 8 months
  Other Names: Diovan
  Arms: Valsartan
Drug: Hydrochlorothiazide — Hydrochlorothiazide 25mg PO daily for 8 months
  Other Names: HCTZ
  Arms: Hydrochlorothiazide

SUMMARY:
Traditionally, obesity is considered an indirect cause of heart disease. Obese individuals typically present with a number of traditional Framingham risk factors (hypertension, dyslipidemia, and type 2 diabetes), predisposing them to heart attacks and subsequent heart failure. However, an emerging body of basic research revisits a hypothesis that fat is a direct cardiotoxin. Under healthy conditions, most triglyceride is stored in fatty tissue (adipocytes) while the amount of triglyceride stored in non-adipocyte tissues (such as the pancreas, the liver, skeletal muscle, and heart) is minimal and very tightly regulated. When this regulation is disrupted, intracellular triglyceride accumulates excessively in these organs ("steatosis") and has been implicated in activating adverse pathways which culminate in irreversible cell death ("lipotoxicity"), leading to several well-recognized clinical syndromes. These include non-alcoholic steatohepatitis (NASH), pancreatic beta-cell failure in type 2 diabetes, and dilated cardiomyopathy.

It has been recently observed that angiotensin II receptor blockers (ARBs) in addition to lowering blood pressure improve insulin sensitivity and decrease the risk for type 2 diabetes. This study will test the above theory in two study groups: Valsartan vs. Hydrochlorothiazide. We hypothesize that in obese humans with elevated myocardial triglycerides, blockade of the renin-angiotensin system (Valsartan group) will reduce myocardial fat with improvement of insulin sensitivity and heart function.

DETAILED DESCRIPTION:
Basic science in animal models of genetic obesity have demonstrated that obese, insulin resistant animals have fatty hearts with reduced functional ability. More importantly, insulin sensitizing treatment of prediabetic rats delayed development of diabetes and improved heart function. A primary aim of our laboratory is to translate basic animal research, suggesting that excessive lipid accumulation in the myocardium is toxic, into the clinical setting using cardiac magnetic resonance imaging/spectroscopy technology. The results of this research may identify new biomarkers and drug targets to prevent cardiac disease in obese humans.

We used our novel in vivo magnetic resonance imaging and spectroscopy technique that enables quantification of triglyceride in human myocardium non-invasively, to demonstrate that obese humans like obese animals are characterized by elevated fat in myocardium. We hypothesize that in obese humans with elevated myocardial TG, blockade of the renin-angiotensin system will reduce myocardial fat with improvement of insulin sensitivity and heart function.

The aims of this study are to test if in obese people with impaired glucose tolerance (IGT):

Aim 1) Valsartan treatment will reduce myocardial fat and will improve heart geometry and function,

Aim 2) therapy with thiazide diuretic hydrochlorothiazide (HCTZ) treatment will elevate myocardial fat.

We are planning to test the action of Valsartan versus HCTZ as we expect that these drugs cause opposite metabolic effects. The landmark trial ALLHAT (Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial) has refocused attention to the thiazide-type diuretics as the first-line therapy for most patients with hypertension. Despite proven reduction in cardiovascular outcomes and low costs, there is on-going concern that one of the major side effect of the thiazides-glucose intolerance-may fuel the current U.S. epidemic of type 2 diabetes. Despite of efficacy and low cost thiazide diuretics are long known to cause insulin resistance, impaired glucose tolerance, and precipitation of overt diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Prediabetic individuals with impaired glucose tolerance (2 hr postprandial glucose > 140mg/dL) or having 3 of 5 Metabolic Syndrome criteria:

  1. Fasting glucose > 100mg/dL;
  2. Waist circumference: men > 102cm, women > 88cm (confirmed with abdominal MRI);
  3. HDL: men < 40mg/dL, women < 50mg/dL;
  4. Triglycerides > 150mg/dL;
  5. Blood pressure > 130/80mmHg;
* Elevated hepatic triglycerides (>5.5%) and myocardial triglycerides (>0.6%)
* Elevated blood triglycerides >150mg/dL
* Age < 50 years

Exclusion Criteria:

* Type 2 Diabetes mellitus
* Prior exposure to renin system blockers or HCTZ
* BP > 160/100mmHg
* Claustrophobia
* Metallic implants in body
* Pregnant or planning to become pregnant
* Prior exposure to statin medications

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2007-08; Primary Completion 2009-08 (Estimated); Study Completion 2009-08 (Estimated)

PRIMARY OUTCOMES:
Myocardial triglyceride levels | 8 months

SECONDARY OUTCOMES:
Hepatic triglyceride levels, insulin sensitivity, abdominal fat mass | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G Victor, MD, Principal Investigator — University of Texas Southwestern Medical Center; Lidia S Szczepaniak, PhD, Study Director — University of Texas Southwestern Medical Center
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States